CLINICAL TRIAL: NCT01732705
Title: Effect of High Intensity Interval Training (HIT) on Insulin Sensitivity in Patients With Type 2 Diabetes
Brief Title: High Intensity Interval Training (HIT) in Patients With Type 2 Diabetes
Acronym: HIT_T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, Flemming Dela, Professor, MD., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIT-T2DM
Record Dates: First submitted 2012-10-12; First posted 2012-11-26 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Insulin sensitivity; High intensity interval training
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HIT (trained leg) DM (Experimental): High intensity interval training for one leg (trained leg) (randomized) in patient with type 2 diabetes
  Interventions: Behavioral: High intensity interval training
- Control leg, DM (No Intervention): Control leg (untrained leg)in patient with type 2 diabetes
- HIT (trained leg), Control subject (Experimental): High intensity interval training for one leg (trained leg) (randomized) in control subject
  Interventions: Behavioral: High intensity interval training
- Control leg, Control subject (No Intervention): Control leg (untrained leg)in control subject

INTERVENTIONS:
Behavioral: High intensity interval training — HIT will be conducted as 2 weeks of one legged high intense interval training (8 sessions every 2nd day). Each training session will consist of 10 x 1 min intervals on ergometer bicycle interspersed with 1 min recovery.
  Other Names: High intense interval training; HIT; HIIT
  Arms: HIT (trained leg) DM; HIT (trained leg), Control subject

SUMMARY:
The purpose of this study is to determine the effect of High Intensity Interval Training (HIT) on insulin sensitivity in skeletal muscle in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Physical exercise increases insulin sensitivity in skeletal muscle in healthy as well as in individuals with type 2 diabetes, but implies a considerable time commitment. High intensity interval training (HIT) is time-efficient exercise consisting of repeated bouts of short duration high intensive workloads. The aim of this study is to determine the effect of HIT in patients with type 2 diabetes, and to clarify the mechanisms of a possible positive effect of HIT.

Exercise is performed as 2 weeks one-legged training on an ergometer bicycle. Thus one leg serves as a control leg. Insulin sensitivity in trained and non-trained muscle will be measured after completion of the overall training program by euglycemic hyperinsulinemic clamp method and a-v catheterization of both legs. Muscle biopsies will be obtained during training period for measuring of muscle glycogen content, and muscle biopsies for further analysis obtained during the experimental day.

ELIGIBILITY:
Inclusion Criteria:

* 10 subjects with Type 2 diabetes. 10 healthy control subjects.
* BMI 28-35
* diet or tablet treatment for diabetes

Exclusion Criteria:

* regular physical activity
* diseases other than type 2 diabetes
* insulin treatment

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 days after last training session (day 17)
  Insulin sensitivity in trained and non-trained muscle will be measured by euglycemic hyperinsulinemic clamp method and a-v catheterization of both legs.

OTHER OUTCOMES:
Glycogen content in skeletal muscle | 17 days. Before and after training session day 1, 7 and 15. Before and immediately after isoglycemic, hyperinsulinemic clamp day 17.
  Analysis of glycogen content from muscle biopsies taken during the training period.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, MD. Prof., Principal Investigator — Xlab, Department of Biomedical Sciences, University of Copenhagen
Locations (1):
- Xlab, Department of Biomedical Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Dela F, Ingersen A, Andersen NB, Nielsen MB, Petersen HHH, Hansen CN, Larsen S, Wojtaszewski J, Helge JW. Effects of one-legged high-intensity interval training on insulin-mediated skeletal muscle glucose homeostasis in patients with type 2 diabetes. Acta Physiol (Oxf). 2019 Jun;226(2):e13245. doi: 10.1111/apha.13245. Epub 2019 Feb 14. PMID 30585698